CLINICAL TRIAL: NCT07165314
Title: Assessment of Provider Position for Prehospital Tracheal Intubation Using Direct Laryngoscopy: Randomized Controlled Trial
Brief Title: Assessment of Provider Position for Prehospital Tracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Cédric Cibotto, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Req-2025-01129
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Tracheal Intubation
Keywords: advanced airway management; laryngoscopy; sitting position; prehospital; manikin; randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free positioning (Active Comparator)
  Interventions: Procedure: Free positioning
- Sitting cross-legged ("Lotus" position) (Experimental)
  Interventions: Procedure: Sitting cross-legged ("Lotus" position)

INTERVENTIONS:
Procedure: Free positioning — Participants are not given instructions on how to position for intubation using direct laryngoscopy.
  Arms: Free positioning
Procedure: Sitting cross-legged ("Lotus" position) — Participants are requested to sit cross-legged for intubation using direct laryngoscopy.
  Arms: Sitting cross-legged ("Lotus" position)

SUMMARY:
Endotracheal intubation may be needed in critically ill patients in the prehospital setting, where difficult conditions may be encountered. The patient may be lying on the ground, thus complicating direct laryngoscopy as the operator's visual axis cannot be properly aligned with the patient's oral-pharyngeal-tracheal axis. The posture sitting cross-legged ("Lotus" position) at the head of the patient may allow an easier alignment of the visual axes due to a lower operator's head position and more stability. We compared the impact of the "Lotus" position with free positioning of the operator for direct laryngoscopy on intubation first pass success rate among novice operators.

ELIGIBILITY:
Inclusion Criteria:

* All resident doctors with 1 to 6 years of post-graduate experience working in the Emergency Department (ED) at Geneva University Hospitals (Hôpitaux Universitaires de Genève (HUG)) and penultimate year of medical school students (5th year) studying at University of Geneva Faculty of Medicine (UGFM) - Performed less than 10 ETIs prior to take part in the research

Exclusion Criteria:

* More than 6 years of post-graduate experience
* Performed more than 10 ETIs prior to take part in the research

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
First Pass Success rate | Periprocedural
  In percentage, defined as achieving successful ETI on the initial attempt. An ETI attempt was counted since the laryngoscope blade was inserted at the dental arch, regardless of whether tracheal tube placement was attempted or not. ETI was considered successful when adequate ventilation was confirmed by chest elevation. The number of intubation attempts were limited to three, with a time limit of 60 seconds allowed per attempt.

SECONDARY OUTCOMES:
Time to Intubation | Periprocedural
  Time in seconds from blade insertion at the dental arch to successful ventilation. A maximum of 60 seconds was allowed per ETI attempt.
Time to Intubation for the first intubation attempt alone | Periprocedural
  Time in seconds from blade insertion at the dental arch to adequate ventilation, ruling out first-attempt failures. A maximum of 60 seconds was allowed per ETI attempt.
Number of intubations attempts | Periprocedural
  An ETI attempt was counted since the laryngoscope blade was inserted at the dental arch, regardless of whether tracheal tube placement was attempted or not. ETI was considered successful when adequate ventilation was confirmed by chest elevation. The number of intubation attempts were limited to three, with a time limit of 60 seconds allowed per attempt.
Cormack and Lehane (CL) score | Periprocedural
  For each attempt, the view of the larynx was assessed by the participant using the Cormack-Lehane score.
Percentage Of Glottis Opening (POGO) score | Periprocedural
  For each attempt, the percentage of glottis opening was assessed by the participant, using the POGO score.
Subjective assessments | Periprocedural
  Perceived difficulty was appraised using a 5-point Likert scale ranging from "Totally Agree" to "Totally Disagree".

CONTACTS AND LOCATIONS:
Overall Officials: Laurent SUPPAN, PD Dr, Study Director — University Hospital, Geneva
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva, Switzerland